CLINICAL TRIAL: NCT04711382
Title: The Use of Faster Acting Aspart in Type 1 Diabetes Patients: Multi-centre Real-world Experience
Brief Title: The Use of Faster Acting Aspart in Type 1 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: Fiasp real-world data
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes; Insulin; Time in Range
Keywords: fast acting insulin; glucometrics
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data on switching from traditional mealtime insulins to fast-acting insulin aspart (Fiasp) in routine clinical practice are sparse. The aim was to evaluate the efficacy and safety of switching from traditional mealtime insulin to Fiasp in a "real-world" clinical practice setting in people with type 1 diabetes in Belgium.

DETAILED DESCRIPTION:
The primary endpoint was the evolution of time in range (TIR, 70-180 mg/dl) at 6 and 12 months. Secondary endpoints included change in HbA1c, BMI, insulin doses, time below range (T<70 and T<54 mg/dl) and time above range (T>180 and T>250 mg/dl).

Retrospective analysis Two-center study

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes patients
* Duration of diabetes > 2 years
* Using CGM for > 6 months

Exclusion Criteria:

* Using SMBG
* Pregnancy
* Using glucocorticoids or immunosuppressive agents
* Active oncological problem

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult type 1 diabetes patients, with a duration of diabetes of > 2 years
Sampling Method: Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Time in Range | 12 months
  Time in target range at 12 months

SECONDARY OUTCOMES:
Time in Range | 6 months
  Time in target range at 6 months
Change in HbA1c | 6 months & 12 months
  Change in HbA1c
Change in weight | 6 months & 12 months
  Change in weight
Change in insulin doses | 6 months & 12 months
  Change in insulin doses
Time below range | 6 months & 12 months
  Change in time below range
Time above range | 6 months & 12 months
  Change in time above range
Coefficient of variation | 6 months & 12 months
  Change in coefficient of variation

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium